CLINICAL TRIAL: NCT04599283
Title: Validation of MenHealth Mobile Uroflowmetry Application
Brief Title: BE Technologies Mobile Uroflowmetry Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BE Technologies Inc (Industry)
Collaborators: Urology of Virginia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 00041138
Record Dates: First submitted 2020-10-12; First posted 2020-10-22 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: BPH; BPH With Urinary Obstruction With Other Lower Urinary Tract Symptoms; BPH Without Urinary Obstruction; BPH Without Urinary Obstruction With Other Lower Urinary Tract Symptoms; Lower Urinary Tract Symptoms; Overactive Bladder; Overactive Bladder Syndrome; Urinary Obstruction; Urinary Incontinence, Urge
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Symptomatic (Active Comparator): 1. You have to be a male patient.
  2. You must have a smartphone (iPhone or Android).
  3. You are at least 35 years old and have already been diagnosed with BPH or Overactive Bladder (OAB) condition OR you are presenting at least one of the following BPH / OAB symptoms:
  1. Frequent or urgent need to urinate 2. Increased frequency of urination at night (nocturia) 3. Difficulty starting urination 4. Weak urine stream or a stream that stops and starts 5. Dribbling at the end of urination 6. Inability to completely empty the bladder 7. Experience urge incontinence - the involuntary loss of urine immediately following an urgent need to urinate
  Interventions: Device: MenHealth Uroflowmeter
- Asymptmatic (Active Comparator): 1. You have to be a male patient.
  2. You must have a smartphone (iPhone or Android).
  3. You are at least 18 years old and have not been diagnosed with BPH or OAB, and you are not presenting any of the above symptoms.
  Interventions: Device: MenHealth Uroflowmeter

INTERVENTIONS:
Device: MenHealth Uroflowmeter — MenHealth Uroflowmeter is a mobile application and FDA cleared medical device that analyzes the sound of urine hitting the toilet water when a male urinates and generates voiding data (maximum flow, average flow, and voided volume) and a flow curve. All test results are saved in an automated voiding diary.
  Other Names: MenHealth Mobile Uroflowmeter

SUMMARY:
This research study is studying MenHealth Mobile Uroflowmetry as a diagnostic tool for LUTS (lower urinary tract symptoms), a group of conditions involving the bladder, urinary sphincter, urethra and the prostate.

DETAILED DESCRIPTION:
As men age, they are at higher risk of developing lower urinary tract symptoms. The cause or source of these symptoms can range from overactive bladder (OAB), urethral stricture disease, and benign prostatic hyperplasia (BPH).

Patients are also often asked to return to clinic to perform a uroflow test in order to:

1. Evaluate for expected post surgical improvement in flow or
2. To investigate the urinary flow in men with new lower urinary tract complaints.

The in-office uroflow test involves an office visit, which often requires a patient copay and other health care resources. In addition, it is performed in an artificial "high pressure" environment and many patients find it difficult to present with a full bladder due to their lower urinary tract symptoms.

This research may help us determine whether an "at home" uroflow test can be used to obtain similar diagnostic data in the patient's natural environment, without the need for an in-office visit. A patient's test results taken at home in a comfortable environment could be reliable and informative for both the patient and the doctor. This data can then be used to determine the appropriate management.

The purpose of this research study is to conduct a performance validation of MenHealth Uroflowmetry application by comparing data obtained by MenHealth Uroflowmetry application with the data obtained by a standard office Uroflowmeter.

The study is investigational. Its goal is to study and compare test results obtained by the study subject using MenHealth application with the test results obtained from the subject's office uroflow test.

About 60 subjects will participate in this study. The 60 subjects will comprise two groups: Group 1/Symptomatic (45 subjects) and Group 2/Asymptomatic (15 subjects).

Subject participation in this study will last approximately 2 weeks and will include 2 study visits to the study center. At the end of the 2 week period, subjects should have a minimum of 10 reliable uroflowmetry tests done at home.

ELIGIBILITY:
Inclusion Criteria:

* You have to be a male patient.
* You must have a smartphone (iPhone or Android).
* For Group 1 (Symptomatic), you are at least 35 years old and have already been diagnosed with BPH or Overactive Bladder (OAB) condition OR you are presenting at least one of the following BPH / OAB symptoms: frequent or urgent need to urinate, increased frequency of urination at night (nocturia), difficulty starting urination, weak urine stream or a stream that stops and starts, dribbling at the end of urination, inability to completely empty the bladder, experience urge incontinence - the involuntary loss of urine immediately following an urgent need to urinate.
* For Group 2 (Asymptomatic), you are at least 18 years old and have not been diagnosed with BPH or OAB, and you are not presenting any of the above symptoms.

Exclusion Criteria:

* Male younger than 18 or older than 90
* Female

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 54 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
MenHealth Uroflowmetry application performance | 2 weeks
  To validate the performance of MenHealth Uroflowmetry application by measuring maximum flow, average flow, and voided volume obtained by MenHealth Uroflowmetry application and comparing this data with corresponding data obtained by a standard office Uroflowmeter. Every individual Uroflowmetry test contains these three parameters ( maximum flow, voided volume, and average flow) as an outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Schultz, MD, Principal Investigator — Urology of Virginia
Locations (1):
- Urology of Virginia, Virginia Beach, Virginia, United States

IPD SHARING:
Plan to Share IPD: No